CLINICAL TRIAL: NCT01424475
Title: LRRK2 Mutation and Parkinson's Disease: A Functional Neuroimaging and Behavioural Study Characterising the Neurocognitive Phenotype
Brief Title: LRRK2 Mutation and Parkinson's Disease
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Following extensive efforts to increase recruitment, it will not be possible to complete the study protocol within a reasonable time
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 114500
Record Dates: First submitted 2011-06-23; First posted 2011-08-29 (Estimated); Last update posted 2017-05-11 (Actual); Status verified 2017-05

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- PKD Patients (Other): PKD Patients with LRRK2 mutation
  Interventions: Genetic: PKD Patients
- Healthy Controls (Other): Healthy Controls with no LRRK2 mutation
  Interventions: Genetic: Healthy

INTERVENTIONS:
Genetic: Healthy — Healthy Volunteers
  Arms: Healthy Controls
Genetic: PKD Patients — PKS Patients
  Arms: PKD Patients

SUMMARY:
The Leucine-Rich Repeat Kinase 2 (LRRK2) is implicated in autosomal dominant Parkinson's disease (PKD). An inhibitor for the leucine-rich repeat kinase 2 (LRRK2) is in pre-clinical development for potential use in treating Parkinson's disease. Patients with PKD have cognitive impairments which develop alongside the typical motor symptoms but a full characterisation of the neurocognitive phenotype of PKD patients with LRRK2 mutation is currently lacking. This observational study conducted on a single visit will assess the phenotypic neurocognitive abnormalities of PKD patients with the LRRK2 mutation with the aim of identifying potential PD endpoints related to the LRRK2 mutation for future Phase I or II clinical trials of LRRK2 inhibitors.

DETAILED DESCRIPTION:
The Leucine-Rich Repeat Kinase 2 (LRRK2) is implicated in autosomal dominant Parkinson's disease (PKD). An inhibitor for the leucine-rich repeat kinase 2 (LRRK2) is in pre-clinical development for potential use in treating Parkinson's disease. Patients with PKD have cognitive impairments which develop alongside the typical motor symptoms but a full characterisation of the neurocognitive phenotype of PKD patients with LRRK2 mutation is currently lacking. This observational study conducted on a single visit will assess the phenotypic neurocognitive abnormalities of PKD patients with the LRRK2 mutation with the aim of identifying potential PD endpoints related to the LRRK2 mutation for future Phase I or II clinical trials of LRRK2 inhibitors.

Approximately 20 subjects with PKD bearing one of the known LRRK2 mutations will be investigated. Approximately 20 healthy subjects without the LRRK2 mutation who are matched with PKD patients will also be evaluated.

Healthy subjects are not expected to be taking medications for PKD. Subjects with PKD may continue their medications for PKD treatment throughout the study, Testing will take place within 30 days of screening, depending on the subject's availability.

ELIGIBILITY:
Any Subject:

Inclusion Criteria:

* Male or female, age: >18 years.
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.
* Sufficiently fluent in English that they are able to understand written and spoken instructions in the opinion of the investigator.

Exclusion Criteria:

* Subjects with previous or current drug or alcohol dependence within 2 years of screening.
* Subjects who are unable to tolerate study procedures including MRI, or who are unable to perform the study procedures (e.g. due to severe musculoskeletal disease).
* Use of other prescription or non-prescription centrally acting drugs, including herbal (eg khat) and dietary supplements within 7 days or 5 half-lives (whichever is longer) prior to the procedures of Day 1, unless in the opinion of the Investigator and GSK Medical Monitor the medication will not interfere with the study procedures or compromise subject safety.
* Pregnant females as determined by positive serum or urine hCG test at screening.
* Lactating females.
* Unwillingness or inability to follow the procedures outlined in the protocol.
* Subject is mentally or legally incapacitated.
* Subject meets any of the MRI exclusion criteria.
* Subject is left-handed.

PKD Patients:

Inclusion Criteria:

* Diagnosis of Parkinson's disease according to the following criteria derived from the UKPD Society brain bank diagnostic criteria for PD (Hughes AJ et al., 1992):

  a) Bradykinesia must be present b) At least one of the following: muscular rigidity Resting tremor postural instability not caused by primary visual, vestibular, cerebellar or proprioceptive dysfunction c) Supportive prospective positive criteria for Parkinson's Disease (three of the following required for definite diagnosis): Resting tremor unilateral onset progressive disorder in first 5 years following onset, persistent asymmetry affecting side on which symptoms first appeared excellent response (70-100%) to levodopa in the clinical judgement of the investigator, based on the medical notes or during standard care d) None of the following clinical features which suggest a diagnosis other than Parkinson's disease: History of repeated strokes with stepwise symptom progression History of repeated head injury History of definite encephalitis Neuroleptic treatment at symptom onset Sustained remission Strictly unilateral features after 3 years Supranuclear gaze palsy Cerebellar signs In first five years following onset, early severe autonomic involvement such as orthostatic hypotension, impotence and bladder dysfunction Early (within 2 years on symptom onset) severe dementia with disturbed memory, language, praxis Babinski sign CT/MRI scan evidence of tumour or hydrocephalus Negative response to 1000mg of levodopa daily in divided doses.

  1-methyl-4-phenyl-1,2,3,6-tetrahydropyridine (MPTP) exposure
* Parkinson's disease in Hoehn & Yahr criteria Stages I-III.
* Confirmed ascertainment as having the G2019S mutation in the LRRK2 gene.

Exclusion Criteria:

* Subjects with clinically significant condition(s) other than Parkinson's disease which, in the opinion of the investigator, would render the subject unsuitable for the study (e.g. psychiatric, haematological, renal, hepatic, endocrinology, neurological [other than Parkinson's disease], cardiovascular, or active malignancy [other than benign skin malignancies]).
* Subjects with prior or current major psychosis (e.g. schizophrenia or psychotic depression) as assessed by the MINI neuropsychiatric interview.
* Subjects with severe clinical dementia as measured by UPDRS.
* Patients who are on centrally acting anti-cholinergic medication that is likely to impair cognitive function.
* Patients with positive drug screen results may still be included at the discretion of the investigator following a discussion of the result with the subject, and following a discussion with the sponsor.

Healthy Subjects (Controls):

Inclusion Criteria:

* Matched to patients with LRRK2 mutation for age, gender, premorbid reading IQ, handedness and smoking status (number of cigarettes smoked per day (0-10, 11-20, 21-30 or 30+)).
* None of the clinical symptoms or signs of Parkinson's disease listed in section 5.2.2.1.
* No family history of more than one first-degree relative with Parkinson's disease to suggest that the subject may be a carrier of one of the genetic mutations of Parkinson's disease.
* Confirmed ascertainment as not having LRRK2 mutation.
* Subject is not a genetically-related family member of a subject with LRRK2 mutation recruited into this study as per criteria above.
* Subject is healthy as determined by a responsible and experienced physician, based on a medical evaluation including medical history, physical examination, laboratory tests and cardiac monitoring. A subject with a clinical abnormality or laboratory parameters outside the reference range for the population being studied may be included only if the Investigator and the GSK Medical Monitor agree that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures.
* No current or past history of Axis I psychiatric disorders as determined by MINI interview.

Exclusion Criteria:

* A positive pre-study drug/alcohol screen.
* Currently taking any prescription medication, in particular medication with a central mechanism of action, unless in the opinion of the Investigator and GSK Medical Monitor the medication will not interfere with the study procedures or compromise subject safety.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2011-08-11 (Actual); Primary Completion 2015-01-12 (Actual); Study Completion 2015-01-12 (Actual)

PRIMARY OUTCOMES:
Imaging (fMRI) | Day 1
  Action Selection, Tower of London, Shape manipulation, Emotional processing
Cognition | Day 1
  Mini Mental State Examination (MMSE), Reward/punishment learning score, Task-set switching, Attentional set-shifting score, Spatial working memory score
Olfactory | Day 1
  Sniffin' sticks
Motor / Other | Day 1
  Unified Parkinson's Disease Rating Scale (UPDRS), Beck Depression Inventory (BDI), Parkinson's Disease Sleep Scale (PDSS), Nonmotor Symptoms Questionnaire, Questionnaire for Impulsive-Compulsive Disorders in Parkinson's Disease, Caffeine/Smoking Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Cambridge, United Kingdom

REFERENCES:
- See also: Results for study 114500 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/114500?search=study&search_terms=114500#rs